CLINICAL TRIAL: NCT06587295
Title: A Phase 1, Open-Label, Dose Escalation and Expansion Study of Intramuscular ACM-CpG Monotherapy in Patients With Advanced/Metastatic Solid Tumors With Prior Response to Immunotherapy Alone or in Combination With Chemotherapy
Brief Title: Intramuscular ACM-CpG Monotherapy in Patients With Advanced/Metastatic Solid Tumors With Prior Response to Immunotherapy Alone or in Combination With Chemotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: ACM Biolabs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACMBxNCCS001
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: ACM-CpG
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escalation (Experimental)
  Interventions: Drug: Intramuscular ACM-CpG Monotherapy (Escalation)
- Expansion (Experimental)
  Interventions: Drug: Intramuscular ACM-CpG Monotherapy (Expansion)

INTERVENTIONS:
Drug: Intramuscular ACM-CpG Monotherapy (Escalation) — Dose escalation for ACM-CpG monotherapy administered via intramuscular injection will similarly be conducted using traditional 3+3 dose escalation. Three dose levels have been planned. If the patient experiences a DLT or two Grade ≥ 2 drug-related toxicity, the dose level will be expanded according to a 3+3 design. The safety and tolerability of each dose level will be assessed by the study team after all patients enrolled in the dose level have been followed for at least 21 days after the first dose of the ACM-CpG (DLT observation period). Once the MTD is reached, the RP2D will be determined.
  Arms: Escalation
Drug: Intramuscular ACM-CpG Monotherapy (Expansion) — Patients will be administered ACM-CpG monotherapy at a dose determined in the dose escalation phase.
  Arms: Expansion

SUMMARY:
ACM-CpG is a CpG-B TLR9 agonist, which in animal models has led to shrinkage and complete disappearance of injected tumors, durable antitumor memory, and growth inhibitory effects on non-injected tumors while intramuscular administration led to durable control of tumors. This Phase I trial will assess the safety and early signs of efficacy of intramuscular injection of ACM-CpG in patients with advanced malignant solid tumors.

The overall objectives of this trial are to establish the safety ACM-CpG.

DETAILED DESCRIPTION:
This is a phase 1, open-label, dose escalation and expansion study of intramuscular ACM-CpG monotherapy in patients with advanced or metastatic solid tumours. Dose escalation will be conducted and the RP2D will be determined for ACM-CpG monotherapy for intramuscular routes of administration. The study will enroll patients who have received prior immunotherapy as standard of care treatment and have had demonstrable radiological responses.

Dose escalation for ACM-CpG monotherapy administered via intramuscular injection will similarly be conducted using traditional 3+3 dose escalation. Three dose levels have been planned. If the patient experiences a DLT or two Grade ≥ 2 drug-related toxicity, the dose level will be expanded according to a 3+3 design.

The safety and tolerability of each dose level will be assessed by the study team after all patients enrolled in the dose level have been followed for at least 21 days after the first dose of the ACM-CpG (DLT observation period). Once the MTD is reached, the RP2D will be determined. The RP2D will be defined based on the observation of MTD in a dose level cohort, to include dose levels below the MTD, or intermediate between the pre-specified dose levels based on an overall assessment of all safety data, as well as all available PK and pharmacodynamic data, and documented objective response observations. RP2D will be a pharmacologically active dose, declared based on an aggregate of multiple factors including PK data evaluating the safety margin based on CpG7909 plasma concentrations across a range of dosing levels compared to prior data (https://pubmed.ncbi.nlm.nih.gov/17696823/) and clinical results.

Dose escalation and expansion will be performed in patients that have previously responded to immune checkpoint therapy alone or in combination with chemotherapy and who have already received standard of care treatment. Following the determination of the RP2D, dose expansion will be performed.

Approximately up to 30 to 40 patients will be enrolled on study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 21 years of age at the time of informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 with no functional deterioration over the previous 2 weeks.
3. Estimated life expectancy of more than 12 weeks.
4. Patients with terminal, Stage 4, advanced or metastatic solid tumors, confirmed histologically or pathologically documented, and who have previously received and clinically responded to ICI alone or in combination chemotherapy with best response by RECIST 1.1 being complete response (CR), partial response (PR) or stable disease (SD) who now have progression of disease and have previously received existing standard of care treatment.
5. Adequate hematologic function, defined by the following:

   1. Absolute neutrophil count (ANC) ≥ 1.5 ×10**9/L, without the use of granulocyte colony stimulating factor such as filgrastim within 2 weeks prior to study treatment.
   2. Platelet count ≥ 100 × 10**9/L without transfusion within 2 weeks (≤ 14 days) prior to study treatment.
   3. Hemoglobin ≥ 9 g/dL without transfusion or erythropoietin within 2 weeks (≤ 14 days) prior to study treatment.
6. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN), and total bilirubin ≤ 5 × ULN. Exception: Patients who have serum bilirubin increases due to documented underlying Gilbert's Syndrome or familial benign unconjugated hyperbilirubinemia. Known Hepatitis B and Hepatitis C carriers are eligible if their liver function falls within specifications stipulated here and for Hepatitis B carriers (HBsAg positive) have low HBV DNA, and for Hepatitis C carriers are HCV RNA negative, as well as having adequate disease control on antiviral therapy as required having commenced at least 1 month prior to enrolment.
7. Adequate renal function defined by either a creatinine clearance ≥ 30 mL/min (by Cockcroft- Gault formula) or serum creatinine (SCr) < 1.5 × ULN
8. Coagulation tests, defined by the following:

   1. Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
   2. International normalized ratio (INR) ≤ 1.5 × ULN. Exception: INR 2 to ≤ 3 × ULN is acceptable for patients on Warfarin anticoagulation.
9. Previous antitumor therapy (including endocrine, chemoradiotherapy/ radiotherapy, targeted therapy, or immunotherapy) stopped at least 4 weeks/5 half lives (whichever is shorter) prior to administration of ACM-CpG. Focal radiation therapy for symptom relief must have been completed at least 2 weeks prior to the first dose of ACM-CpG.
10. Previous AEs including irAE, have been improved to baseline or Grade ≤ 1 NCI CTCAE v5.0 (except for patients with alopecia, neuropathy, now or other AEs deemed to be G2 but clinically well managed), and specifically prior immune-related adverse events (irAEs) controlled and improved back to baseline or to Grade ≤ 2 NCI CTCAE v5.0, for example ICI related hypothyroidism requiring repletion with thyroid hormone.
11. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test positive is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 26 weeks after the last dose of the study medication.
12. Male subjects should agree to use adequate method of contraception starting with the first dose of study therapy through 26 weeks after the last dose of the study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Patients receiving granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), erythropoietin, or blood (red blood cell [RBC] or platelet) transfusion within 14 days prior to the first dose of the study drug.
2. Any uncontrolled active infections requiring systemic antimicrobial treatment (viral, bacterial, or other), or uncontrolled or poorly controlled diabetes as evidenced by screening (baseline) Hb1Ac ≥7.5, asthma, chronic obstructive pulmonary disease (COPD).
3. Known positive test result for human immunodeficiency virus (HIV) (except the disease is clinically controlled) or acquired immune deficiency syndrome (AIDS).
4. Patients with any type of primary immunodeficiency or autoimmune disorder requiring treatment.
5. Major surgery within 4 weeks prior to the first dose of the study drug.
6. Pregnant or nursing
7. Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC)/bone marrow (BM) transplantation.
8. Clinically significant cardiac conditions, including myocardial infarction within the last 6 months, uncontrolled angina, viral myocarditis, pericarditis, cerebrovascular accident, or other acute uncontrolled heart disease < 3 months prior to the first dose of the study drug.
9. Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose of study drug.
10. Live viral vaccine therapies within 4 weeks prior to the first dose of study drug.
11. Any known, documented, or suspected history of illicit substance abuse.
12. Any other disease or clinically significant abnormality in laboratory parameters, including serious medical or psychiatric illness/condition, which in the judgment of the Investigator might compromise the safety of the patient or integrity of the study, interfere with the patient participation in the trial or compromise the trial objectives.
13. Patients with systemic disease requiring systemic pharmacologic doses of corticosteroids greater than 10 mg daily prednisolone (or equivalent) are excluded

    * Subjects who are currently receiving steroids at a dose of <= 10 mg daily do not need to discontinue steroids prior to enrollment.
    * Subjects that require topical, ophthalmological, and inhalational steroids would not be excluded from the study.
    * Subjects who require active immunosuppression of greater than the steroid dose discussed above for any reason are excluded.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days (1 cycle)
  Highest dose level at which less than one-third of the patients in the dose level experienced dose limiting toxicities (DLTs) during the first cycle of treatment.
Recommended phase 2 dose (RP2D) | Up to 2 years.
  To be determined based on the MTD or the totality of the safety and efficacy data if the MTD is not reached.
Safety of ACM-CpG Monotherapy | Up to 2 years.
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), including changes in laboratory parameters.
Tolerability of ACM-CpG Monotherapy | Up to 2 years.
  In terms of dose interruptions, reductions and dose intensity.
Incidence of antibody development against PEG | Up to 2 years.
Correlations of antibody development against PEG with incidence of AEs | Up to 2 years.
Correlations of antibody development against PEG with severity of AEs | Up to 2 years.
Correlations of antibody development against PEG with objective response rate (ORR) | Up to 2 years.
Objective response rate (ORR) | Up to 2 years.
  Percentage of patients with best overall response of Complete Response or Partial Response, in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST). Summarized by dose level.
Disease control rate (DCR) | Up to 2 years.
  Percentage of patients with best overall response of Complete Response or Partial Response or Stable Disease, in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST). Summarized by dose level.
Duration of response (DOR) | Up to 2 years.
  The time from the earliest date of documented Complete Response or Partial Response, in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune RECIST (iRECIST), until documented disease progression or death (by any cause, in the absence of progression), among the subset of patients who achieve Complete Response or Partial Response. In progression-free patients, DOR will be censored at the time of the last evaluable tumor assessment following the earliest date of documented Complete Response or Partial Response.
Progression-free survival (PFS) | Up to 2 years.
  The time from first study treatment until documented disease progression or death (by any cause, in the absence of progression). In progression-free patients, PFS will be censored at the time of the last evaluable tumor assessment (RECIST v1.1 and iRECIST).
Overall survival (OS) | Up to 2 years.
  The time from first study treatment to death due to any cause. Patients alive or lost to follow-up will be censored at the last date known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Amit Jain, MBBS, MRCP (UK), MMed, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No